CLINICAL TRIAL: NCT04510051
Title: Phase I Study of Cellular Immunotherapy Using Memory Enriched T Cells Lentivirally Transduced to Express an IL13Rα2-Targeting, Hinge-Optimized, 41BB-Costimulatory Chimeric Receptor and a Truncated CD19 for Children With Recurrent/Refractory Malignant Brain Tumors
Brief Title: CAR T Cells After Lymphodepletion for the Treatment of IL13Rα2 Positive Recurrent or Refractory Brain Tumors in Children
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19130; NCI-2020-05158 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19130 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Malignant Brain Neoplasm; Recurrent Malignant Brain Neoplasm; Refractory Malignant Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy, IL13(EQ)BBzeta/CD19t+ T cells) (Experimental): Patients receive cyclophosphamide intravenously IV on days -5 and -4, and fludarabine IV on days -5 to -2. Patients then receive autologous IL13(EQ)BBzeta/CD19t+ T cells intraventricularly over 5 minutes QW on day 0. Treatment with autologous IL13(EQ)BBzeta/CD19t+ T cells repeats every 7 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients may receive additional cycles of IL13(EQ)BBzeta/CD19t+ T cells as long as they continue to meet eligibility criteria and have doses available for infusion.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: IL13Ralpha2-specific Hinge-optimized 41BB-co-stimulatory CAR Truncated CD19-expressing Autologous T-Lymphocytes

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Biological: IL13Ralpha2-specific Hinge-optimized 41BB-co-stimulatory CAR Truncated CD19-expressing Autologous T-Lymphocytes — Given intraventricularly
  Other Names: Autologous IL13(EQ)BBzeta/CD19t+ TCM-enriched T Cells

SUMMARY:
This phase I trial investigates the side effects of chemotherapy and cellular immunotherapy in treating children with IL13Ralpha2 positive brain tumors that have come back after a period of improvement (recurrent) or do not respond to treatment (refractory). Cellular immunotherapy (IL13(EQ)BBzeta/CD19t+ T cells) are brain-tumor specific cells that may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as as cyclophosphamide and fludarabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Many patients with brain tumor respond to treatment, but then the tumor starts to grow again. Giving chemotherapy in combination with cellular immunotherapy may kill more tumor cells and improve the outcome of treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the feasibility and safety of lymphodepleting chemotherapy followed by cellular immunotherapy utilizing IL13Ralpha2-specific hinge-optimized 41BB-co-stimulatory chimeric antigen receptor [CAR] truncated CD19-expressing autologous T-lymphocytes (IL13[EQ]BBzeta/CD19t+ Tn/mem cells) administered by intraventricular (ICV) delivery for pediatric participants with IL13Ralpha2+ recurrent/refractory brain tumors.

SECONDARY OBJECTIVES:

I. To describe persistence and expansion of CAR T cells in peripheral blood (PB) and cerebrospinal (CSF).

II. To describe cytokine levels (PB, and CSF) over the study period.

III. In research participants who receive the full schedule of 4 CAR T cell cycles:

IIIa. To estimate 6-month progression free survival (PFS) rate per disease. IIIb. To estimate disease response rates per disease. IIIc. To estimate 1-year overall survival rate per disease. IV. To evaluate the use of circulating tumor deoxyribonucleic acid (ctDNA) to evaluate tumor burden.

V. For study participants who undergo an additional biopsy/resection or autopsy:

Va. To evaluate CAR T cell persistence in the tumor tissue and the location of the CAR T cells with respect to the infusion site. Vb. To evaluate IL13Ralpha2 antigen expression levels on tumor tissue pre and post CAR T cell therapy.

OUTLINE: This is a dose-escalation study of IL13(EQ)BBzeta/CD19t+ T cells.

Patients receive cyclophosphamide intravenously (IV) on days -5 and -4, and fludarabine IV on days -5 to -2. Patients then receive autologous IL13(EQ)BBzeta/CD19t+ T cells intraventricularly over 5 minutes once a week (QW) on day 0. Treatment with autologous IL13(EQ)BBzeta/CD19t+ T cells repeats every 7 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients may receive additional cycles of IL13(EQ)BBzeta/CD19t+ T cells as long as they continue to meet eligibility criteria and have doses available for infusion.

After completion of study treatment, patients are followed for up at 30 days, 3, 6, 9, and 12 months, and then yearly for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies
* Karnofsky Performance Status (KPS) >= 60% except for loss of mobility due to disease involvement; e.g., confinement to a wheelchair due to spinal cord compression
* Life expectancy > 4 weeks
* Participant has a prior histologically-confirmed malignant brain neoplasm and has progressed after prior conventional therapy
* Radiographic evidence of progression/recurrence of the measurable disease more than 12 weeks after the end of the initial conventional therapy (including initial radiation therapy)
* City of Hope (COH) clinical pathology confirms IL13Ralpha2+ tumor expression by immunohistochemistry (IHC) at the initial tumor presentation or recurrent disease (H-score >= 50)
* If the participant has a shunt, it must be programmable and the participant must be able to tolerate the shunt being switched off for at least 2 consecutive days
* Platelets >= 50,000/mm^3 (performed within 6 weeks of signing the main informed consent)
* Total bilirubin =< 2 X upper limit of normal (ULN) (unless has Gilbert's disease) (performed within 6 weeks of signing the main informed consent)
* Aspartate transaminase (AST) =< 2 x ULN (performed within 6 weeks of signing the main informed consent)
* Alanine transferase (ALT) =< 2 x ULN (performed within 6 weeks of signing the main informed consent)
* Creatinine clearance of >= 75mL/min/1.73m^2 (performed within 6 weeks of signing the main informed consent)
* Seronegative for human immunodeficiency virus (HIV) antigen (Ag)/antibody (Ab) combo, hepatitis C virus (HCV)* and active HBV (surface antigen negative) (performed within 6 weeks of signing the main informed consent)

  * If positive, hepatitis C ribonucleic acid (RNA) quantitation must be performed
* Women of childbearing potential (WOCBP): Negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required (to be performed within 6 weeks of signing the main informed consent)
* Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy.

  * Childbearing potential defined as not being surgically sterilized (males and females) or have not been free, once initiated, from menses for > 1 year (females only)
* ELIGIBILITY TO PROCEED WITH PERIPHERAL BLOOD MONONUCLEAR COLLECTION (PBMC) COLLECTION
* Research participant must not require more than 0.1mg/kg/day total dose (0.03mg/kg/dose three times per day, max of 6mg/day) of Dexamethasone on the day of peripheral blood mononuclear cell (PBMC) collection
* Research participant must have appropriate venous access
* At least 2 weeks must have elapsed since the research participant received his/her last dose of prior targeted agents, chemotherapy or radiation
* Note: If a research participant weighs less than 50kgs, the study team should provide the Donor Apheresis Center (DAC) with the participant's current weight so that institutional guidelines can be followed
* ELIGIBILITY TO PROCEED WITH INDWELLING CENTRAL NERVOUS SYSTEM (CNS) CATHETER PLACEMENT
* Serum creatinine < 1.6 mg/dL
* White blood cell (WBC) >= 2,000/dL
* Absolute neutrophil count (ANC) >= 1,000
* Platelets > 50,000/dL
* International normalized ratio =< 1.3
* Bilirubin < 1.5 mg/dL
* Alanine transferase (ALT) and aspartate transaminase (AST) < 2 x upper limits of normal
* KPS >= 60% except for loss of mobility due to disease involvement; e.g., confinement to a wheelchair due to spinal cord compression
* Second-line radiation therapy (post-leukapheresis) completed at least 4 weeks prior to surgical resection or biopsy/catheter placement
* ELIGIBILITY TO PROCEED WITH LYMPHODEPLETION
* Pulmonary: Research participant does not require supplemental oxygen to keep saturation greater than 95% and/or does not have presence of any radiographic abnormalities on chest x-ray that are progressive
* Cardiac: Research participant does not require pressor support and/or does not have symptomatic cardiac arrhythmias
* Active infection: Research participant does not have a fever exceeding 38.5 degree celsius; there is an absence of positive blood cultures for bacteria, fungus, or virus within 48-hours prior to CAR T cell infusion and/or there aren't any indications of meningitis
* Hepatic: Research participant serum total bilirubin or transaminases does not exceed 2 x normal limit
* Renal: Research participant serum creatinine < 1.8 mg/dL
* Neurologic: Research participant does not have uncontrolled seizure activity following surgery prior to starting lymphodepletion
* ELIGIBILITY TO PROCEED WITH EACH CAR T CELL INFUSION
* Research participant has a released cryopreserved T cell product
* Research participant does not require supplemental oxygen to keep saturation greater than 95% and/or does not have presence of any radiographic abnormalities on chest x-ray that are progressive
* Research participant does not require pressor support and/or does not have symptomatic cardiac arrhythmias
* Research participant does not have a fever exceeding 38.5 degree celsius; there is an absence of positive blood cultures for bacteria, fungus, or virus within 48-hours prior to T cell infusion and/or there aren't any indications of meningitis
* Research participant serum total bilirubin or transaminases does not exceed 2 x normal limit
* Research participant serum creatinine < 1.8 mg/dL
* Research participant does not have uncontrolled seizure activity
* Research participant platelet count must be >= 50,000. However, if platelet level is between 25,000-49,000, then T-cell infusion may proceed after platelet transfusion is given and the post transfusion platelet count is >= 50,000
* Research participants must not require more than 0.1mg/kg/day total dose (0.03mg/kg/dose three times per day, max of 6mg/day) of dexamethasone during CAR T cell therapy
* Wash-out requirements:

  * At least 6 weeks since the completion of a nitrosourea-containing chemotherapy regimen;
  * At least 23 days since the completion of temozolomide and/or 4 weeks for any other non-nitrosourea-containing cytotoxic chemotherapy regimen. If a patient's most recent treatment was with a targeted agent only, and s/he has recovered from any toxicity of this targeted agent, then a waiting period of only 2 weeks is needed from the last dose
  * For bevacizumab the wash out period of at least 4 weeks is required before starting study treatment

Exclusion Criteria:

* Pulmonary: Research participant requires supplemental oxygen to keep saturation greater than 95% and the situation is not expected to resolve within 2 weeks
* Cardiac: Research participant requires pressor support and/or has symptomatic cardiac arrhythmias
* Renal: Research participant requires dialysis
* Neurologic: Research participant has uncontrolled seizure activity and/or clinically evident progressive encephalopathy
* Failure of research participant to understand the basic elements of the protocol and/or the risks/benefits of participating in this phase I study. A legal guardian may substitute for the research participant
* Research participant with any non-malignant intercurrent illness which is either poorly controlled with currently available treatment, or which is of such severity that the study team deems it unwise to enter the research participant on protocol shall be ineligible
* Research participant with any other active malignancies
* Research participant being treated for severe infection or recovering from major surgery is ineligible until recovery is deemed complete by the study team
* Research participant with any uncontrolled illness including ongoing or active infection. Research participant with known active hepatitis B or C infection; research participant with any signs or symptoms of active infection, positive blood cultures or radiological evidence of infections
* Research participant who has confirmed HIV positivity within 4 weeks of enrollment
* Females only: Pregnant or breastfeeding
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Ages: 4 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-12-04 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 1 year after the last chimeric antigen response (CAR) T cell infusion
  Will assess the incidence of grade 3 toxicities, dose limiting toxicities, and all other toxicities. Toxicity and adverse events will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 and the revised cytokine release syndrome (CRS) grading system. Symptoms and toxicities will be evaluated by physical exam and blood chemistry/hematology results and adverse event reporting. Rate and associated 90% Clopper and Pearson binomial confidence limits (90% CI) will be estimated for participants experiencing dose limiting toxicities. Tables will be created to summarize all toxicities and side effects by time post treatment, organ, severity and disease subgroup.

SECONDARY OUTCOMES:
Persistence and expansion of CAR T cells | Up to 1 year after the last CAR T cell infusion
  Will assess CAR T cells detected in peripheral blood and cerebrospinal fluid (CSF). Descriptive statistical and graphical methods will be used to describe persistence and expansion of the CAR T cells (peripheral blood [PB] and CSF).
Peripheral blood and CSF cytokine levels | Up to 1 year after the last CAR T cell infusion
  Descriptive statistical and graphical methods will be used to describe cytokine levels (PB and CSF).
Peripheral blood and CSF immune cell characterization | Up to 1 year after the last CAR T cell infusion
Progression free survival | From time of lymphodepletion to the event date (progressionor death), assessed at 6 months
Overall survival | From time of lymphodepletion to date of death, assessed at 1 year after the last CAR T cell infusion
Disease response | Up to 1 year after the last CAR T cell infusion
  Will estimate the rate (90% confidence interval [CI]) of disease response Disease status will be assessed by the grading of the tumor responses performed according to the Response Assessment in Neuro-Oncology Criteria (RANO) criteria.
CAR T cells detected in tumor tissue | Up to 1 year after the last CAR T cell infusion
IL13Ralpha2 antigen expression levels in tumor tissue | Up to 1 year after the last CAR T cell infusion
Circulating tumor deoxyribonucleic acid (ctDNA) assessments | Up to 1 year after the last CAR T cell infusion
  Descriptive statistical and graphical methods will be used to describe ctDNA.

CONTACTS AND LOCATIONS:
Overall Officials: Leo D Wang, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - C.S. Mott Children's Hospital, University of Michigan, Ann Arbor, Michigan